CLINICAL TRIAL: NCT02924246
Title: MOSAIC-2: Effect of Raw Milk on the Immune Response Upon Cholera Vaccination
Brief Title: Effect of Milk on the Vaccination Response
Acronym: MOSAIC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL56906.081.16
Record Dates: First submitted 2016-09-29; First posted 2016-10-05 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2017-01

CONDITIONS: Infection
Keywords: immunity; vaccination; milk
MeSH Terms: conditions — Infections | interventions — Dukoral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (Placebo Comparator): Regular cholera vaccination
  Interventions: Biological: cholera vaccination
- Raw milk (Active Comparator): Cholera vaccination - raw milk
  Interventions: Biological: cholera vaccination; Other: raw milk
- Pasteurized milk (Active Comparator): Cholera vaccination - pasteurized milk
  Interventions: Biological: cholera vaccination; Other: pasteurized milk
- UHT milk (Active Comparator): Cholera vaccination - UHT milk
  Interventions: Biological: cholera vaccination; Other: UHT milk

INTERVENTIONS:
Biological: cholera vaccination — Oral cholera vaccination on day 0 and day 14
  Other Names: Dukoral
Other: raw milk — raw milk
  Arms: Raw milk
Other: pasteurized milk — pasteurized milk
  Arms: Pasteurized milk
Other: UHT milk — UHT milk
  Arms: UHT milk

SUMMARY:
Rationale: Oral vaccination is known to induce a systemic immune response as well as an immune response in mucosal tissues, and can therefore serve as a model to study systemic and mucosal immunity. In this study, the oral cholera vaccine Dukoral® was chosen as model vaccine. The kinetics of the immune response and the interaction with a raw milk matrix have been evaluated in a previous, pilot study (NL49042.081.14). Based on the outcomes of this pilot, in this study oral cholera vaccination will be applied to study the support of immunity by raw milk, compared to heat-treated milk. The study design has been optimised based on previous results: study duration is extended and sample size is based on relevant change and known variation in the primary outcome parameters.

Infections are an important worldwide cause of death, both in elderly and young children. Therefore, support of immunity could help to reduce the incidence of infections. To screen the potential of specific foods or food ingredients to support immunity, oral vaccination can serve as a model. In a previous study, this model was developed using oral cholera vaccination in human adult volunteers. In that study, raw milk was shown to support the immune response to vaccination. In this follow-up study, the effect of raw milk will be compared with pasteurized and ultra-heat treated (UHT) milk.

Objective: To investigate whether pasteurized milk and/or UHT milk are able to enhance the immune response as induced by oral cholera vaccination, in comparison to raw milk and to regular vaccination.

Study design: The study is designed as a single-blind randomized controlled trial of 6 weeks.

Study population: Healthy subjects of 18-50 years of age.

Interventions: 1) Raw milk, obtained from farms that comply to the high quality requirements for production of raw milk, and that has been screened according to the safety criteria for raw milk; 2) commercially available full-fat UHT milk; 3) commercially available full-fat pasteurized milk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 yr
* Signed informed consent
* Availability of internet connection
* Male or female
* Willing to stop blood donation at the blood bank during the study period

Exclusion Criteria:

* Currently participating in another clinical trial
* Previous Cholera, Salmonella, or E. coli vaccination
* Tonsillectomy
* Acute gastroenteritis in the past 2 months
* Use of antibiotics in the past 2 months
* Hypersensitivity to the vaccine, to formaldehyde or to any of the excipients (sodium salts)
* Pregnancy or lactating
* Not willing to drink raw milk
* Allergic to milk or lactose-intolerant
* Disease of GI tract, liver, gall bladder, kidneys, thyroid gland
* Immune-compromised
* Use of immunosuppressive drugs
* Drug abuse, and not willing/able to stop this during the study
* Excessive alcohol usage (men: >4 consumptions/day or >20 consumptions/week; women: >3 consumptions/day or >15 consumptions/week)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in cholera toxin-specific IgA and IgG antibody level in serum as a marker of the vaccination response | baseline and day 14, 28, 42

SECONDARY OUTCOMES:
Change in the cholera toxin-specific IgA and IgG antibody level in nasal wash as a marker of the vaccination response | baseline and day 14, 28, 42
Change in the cholera toxin-specific IgA and IgG antibody level in saliva as a marker of the vaccination response | baseline and day 14, 28, 42
Change in the cholera toxin-specific IgA antibody level in feces as a marker of the vaccination response | baseline and day 14, 28, 42

OTHER OUTCOMES:
Change in the expression of intestinal and mucosal homing markers on IgA and IgG antibody-secreting B cells in peripheral blood, measured by flow cytometry, as markers of the route of modulation of the vaccination response | baseline and day 14
Cholera toxin-specific T cell proliferation as marker of modulation of the vaccination response | baseline and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Els van Hoffen, PhD, Principal Investigator — NIZO Food Research
Locations (1):
- NIZO food research, Ede, Netherlands

IPD SHARING:
Plan to Share IPD: No